CLINICAL TRIAL: NCT05711719
Title: Vericiguat in Patients With Metabolic Syndrome and Coronary Vascular Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00310207
Record Dates: First submitted 2022-12-06; First posted 2023-02-03 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Metabolic Syndrome; Coronary Microvascular Dysfunction
Keywords: Cardiac Magnetic Resonance Imaging
MeSH Terms: conditions — Metabolic Syndrome | interventions — vericiguat

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vericiguat (Experimental): Initial 2.5 mg/day for two weeks, then 5 mg/day for two weeks, and then 10 mg/day for two weeks. Systolic blood pressure will be measured before and following each titration The participant will receive the final titration dose for a total of six weeks.. The drug is administered as an oral tablet once daily.
  Interventions: Drug: Vericiguat
- Placebo (Placebo Comparator): A placebo tablet will be administered orally once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vericiguat — Up-titration will be performed as guided by the evaluation of blood pressure and clinical symptoms
  Other Names: Verquvo
  Arms: Vericiguat
Drug: Placebo — Administered the same way
  Arms: Placebo

SUMMARY:
Coronary vascular dysfunction is one of the "final common pathways" for the impact of multiple cardiovascular risk factors. The investigators will conduct a randomized, double-blind placebo-controlled study in individuals with the metabolic syndrome and baseline coronary vascular dysfunction to evaluate the impact of vericiguat, a stimulator of soluble guanylyl cyclase, on coronary vascular function using non-invasive cardiac magnetic resonance imaging.

DETAILED DESCRIPTION:
Despite advances in medical therapy for the prevention of coronary artery disease, such as the treatments for high blood pressure and elevated cholesterol, several hundred thousand Americans continue to experience heart attacks every year. This may be related to risk factors which are not now identified and therefore treated. Endothelial dysfunction indexes the adverse impact of multiple risk factors and thus provides the opportunity to evaluate the benefit of an intervention which may improve function.

Forty-five participants with metabolic syndrome and coronary vascular dysfunction will be randomized in a 2:1 ratio to receive vericiguat or placebo. Following randomization, the participants will undergo a study drug titration phase as follows: Initial 2.5 mg/day for two weeks, then 5 mg/day for two weeks, and then 10 mg/day for two weeks. This titration protocol is the one stated in the FDA package insert for vericiguat. The vericiguat formulary will be an FDA approved version obtained by the Johns Hopkins Medical Institutions Pharmacy from Merck (manufacturer of vericiguat) and will be maintained by the Johns Hopkins Investigational Drug Service until it is administered.

Cardiac MRI with isometric handgrip exercise, as well as echocardiography and blood studies will be used to assess coronary vascular and cardiac function and biomarkers indicative of nitric oxide pathways and factors impacting that pathway. The same procedures will be repeated at the end of the 6-10 week study drug administration period with an identical protocol, with special attention taken on the MRI to interrogate the same coronary segments as those studied at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age range 35-85 years
* Presence of the metabolic syndrome defined by the National Cholesterol Education Program, Adult Treatment Panel III (NCEP ATP III) definition, with at least three of the following five criteria:

  * waist circumference > 40 inches (men) or >35 inches (women)
  * blood pressure >130/80 mmHg
  * fasting triglyceride (TG) level >150 mg/dL
  * fasting high-density lipoprotein (HDL) cholesterol level <40mg/dL in men or <50mg/dL in women
  * Fasting blood glucose >100 mg/dL, or hemoglobin A1c greater or equal to 5.7%
* Either one of the following:

  * Men ≤ 40 or women ≤ 50 years of age with no history or symptoms of ischemic heart disease, or
  * Men >40 or women >50 years of age with either one of the following

    * a coronary angiography within the past 24 months showing no significant coronary artery disease in a t least one major vessel, defined as >50% stenosis of the left main coronary artery and/or >70% stenosis of another major coronary vessel, or
    * a coronary artery calcium score obtained within the prior 24 months or if no prior calcium scan, one performed as a research study following consent with a Agatston score <10 in at least one major coronary vessel.
* IHE-induced %-change in coronary flow ≤13%

Exclusion Criteria:

* Systolic blood pressure <110 mm Hg
* Current or anticipated use of long-acting nitrates, soluble guanylate cyclase (sGC) stimulators, or phosphodiesterase type 5 (PDE5) inhibitors
* Hematocrit <30%
* Unable to understand the risks, benefits, and alternatives of participation so as to provide informed consent
* Women who are pregnant.
* Women with reproductive capacity not using an acceptable form of contraception
* History of claustrophobia
* Inability to lie flat and still for 45 minutes
* Presence of non-magnetic resonance (MR)-compatible objects or devices, such as intra-orbital debris, intra-auricular implants, intra-cranial clips, an implanted defibrillator or a pacemaker
* History as a machinist, welder, metal worker or a similar activity that poses the risk of metal exposure to the eyes

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten M Leucker, M.D., Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Tsao CW, Aday AW, Almarzooq ZI, Alonso A, Beaton AZ, Bittencourt MS, Boehme AK, Buxton AE, Carson AP, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Ferguson JF, Generoso G, Ho JE, Kalani R, Khan SS, Kissela BM, Knutson KL, Levine DA, Lewis TT, Liu J, Loop MS, Ma J, Mussolino ME, Navaneethan SD, Perak AM, Poudel R, Rezk-Hanna M, Roth GA, Schroeder EB, Shah SH, Thacker EL, VanWagner LB, Virani SS, Voecks JH, Wang NY, Yaffe K, Martin SS. Heart Disease and Stroke Statistics-2022 Update: A Report From the American Heart Association. Circulation. 2022 Feb 22;145(8):e153-e639. doi: 10.1161/CIR.0000000000001052. Epub 2022 Jan 26. PMID 35078371
- [Background] Grundy SM, Brewer HB Jr, Cleeman JI, Smith SC Jr, Lenfant C; American Heart Association; National Heart, Lung, and Blood Institute. Definition of metabolic syndrome: Report of the National Heart, Lung, and Blood Institute/American Heart Association conference on scientific issues related to definition. Circulation. 2004 Jan 27;109(3):433-8. doi: 10.1161/01.CIR.0000111245.75752.C6. No abstract available. PMID 14744958
- [Background] Davignon J, Ganz P. Role of endothelial dysfunction in atherosclerosis. Circulation. 2004 Jun 15;109(23 Suppl 1):III27-32. doi: 10.1161/01.CIR.0000131515.03336.f8. PMID 15198963
- [Background] Hays AG, Iantorno M, Soleimanifard S, Steinberg A, Schar M, Gerstenblith G, Stuber M, Weiss RG. Coronary vasomotor responses to isometric handgrip exercise are primarily mediated by nitric oxide: a noninvasive MRI test of coronary endothelial function. Am J Physiol Heart Circ Physiol. 2015 Jun 1;308(11):H1343-50. doi: 10.1152/ajpheart.00023.2015. Epub 2015 Mar 27. PMID 25820391
- [Background] Hays AG, Hirsch GA, Kelle S, Gerstenblith G, Weiss RG, Stuber M. Noninvasive visualization of coronary artery endothelial function in healthy subjects and in patients with coronary artery disease. J Am Coll Cardiol. 2010 Nov 9;56(20):1657-65. doi: 10.1016/j.jacc.2010.06.036. PMID 21050976
- [Background] Armstrong PW, Roessig L, Patel MJ, Anstrom KJ, Butler J, Voors AA, Lam CSP, Ponikowski P, Temple T, Pieske B, Ezekowitz J, Hernandez AF, Koglin J, O'Connor CM. A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of the Efficacy and Safety of the Oral Soluble Guanylate Cyclase Stimulator: The VICTORIA Trial. JACC Heart Fail. 2018 Feb;6(2):96-104. doi: 10.1016/j.jchf.2017.08.013. Epub 2017 Oct 11. PMID 29032136
- [Background] Jones SP, Bolli R. The ubiquitous role of nitric oxide in cardioprotection. J Mol Cell Cardiol. 2006 Jan;40(1):16-23. doi: 10.1016/j.yjmcc.2005.09.011. Epub 2005 Nov 8. PMID 16288777
- [Background] Tsai EJ, Kass DA. Cyclic GMP signaling in cardiovascular pathophysiology and therapeutics. Pharmacol Ther. 2009 Jun;122(3):216-38. doi: 10.1016/j.pharmthera.2009.02.009. Epub 2009 Mar 21. PMID 19306895
- [Background] Stasch JP, Pacher P, Evgenov OV. Soluble guanylate cyclase as an emerging therapeutic target in cardiopulmonary disease. Circulation. 2011 May 24;123(20):2263-73. doi: 10.1161/CIRCULATIONAHA.110.981738. No abstract available. PMID 21606405

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 45 participants were enrolled (provided written informed consent) and underwent screening MRI. 11 participants were excluded from the study before assignment to veiciguat or placebo: six had normal coronary endothelial function, image quality was poor in two, one experienced claustrophobia, one withdrew and one was lost to follow-up. 34 participants were subsequently randomized.
Period: Overall Study
Arm/Group | Vericiguat | Placebo
Started | 23 | 11
Completed | 21 | 11
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vericiguat | Placebo | Total
Number analyzed (Participants) | 23 | 11 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (8.9) | 59.6 (7.5) | 60.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 16 | 4 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 11 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 18 | 9 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Coronary Cross-sectional Area (in mm²) Within the Vericiguat Group as Assessed by Magnetic Resonance Imaging (MRI)
Description: The difference in absolute change in coronary cross-sectional area (in mm²) from rest to isometric handgrip exercise (IHE) in the group randomized to vericiguat from that measured at baseline, prior to the initiation of vericiguat, to that measured at the end of the study drug administration period, six weeks following initiation of the titrated dose, as assessed by MRI.
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Population: Two participants who were assigned to the Vericiguat group withdrew. One withdrew due to personal bereavement following the unexpected death of a close friend, and the other withdrew due to lightheadedness and nausea following alcohol intake.
Measure: Mean (Standard Deviation); unit: mm^2
Groups:
- Vericiguat (Baseline): Initial 2.5 mg/day for two weeks, then 5 mg/day for two weeks, and then 10 mg/day for two weeks. Systolic blood pressure will be measured before and following each titration The participant will receive the final titration dose for a total of six weeks.. The drug is administered as an oral tablet once daily.
  Vericiguat: Up-titration will be performed as guided by the evaluation of blood pressure and clinical symptoms
- Vericiguat Group (Follow-up Visit): Initial 2.5 mg/day for two weeks, then 5 mg/day for two weeks, and then 10 mg/day for two weeks. Systolic blood pressure will be measured before and following each titration The participant will receive the final titration dose for a total of six weeks.. The drug is administered as an oral tablet once daily.
Arm/Group | Vericiguat (Baseline) | Vericiguat Group (Follow-up Visit)
Number analyzed (Participants) | 21 | 21
mm^2 | -1.11 (1.17) | 0.40 (1.28)
Statistical Analysis 1: Comparison: Vericiguat (Baseline) vs Vericiguat Group (Follow-up Visit); The analysis compares the absolute change in coronary cross-sectional area (mm²) from that at rest to that during isometric handgrip exercise in the Vericiguat group between that measured at baseline and that measured at six weeks following initiation of titrated dose; Test type: Other — Single group analysis; p = 0.0005, t-test, 2 sided

2. Primary Outcome: Relative Change in Coronary Cross-sectional Area (as Percentage) Within the Vericiguat Group as Assessed by Magnetic Resonance Imaging (MRI)
Description: The difference in relative change in coronary cross-sectional area (in %) from rest to isometric handgrip exercise (IHE) in the group randomized to vericiguat from that measured at baseline prior to the initiation of vericiguat, to that measured at the end of the study drug administration period, six weeks following initiation of the titrated dose, as assessed by MRI.
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vericiguat (Baseline) | Vericiguat Group (Follow-up Visit)
Number analyzed (Participants) | 21 | 21
percent change | -6.8 (6.7) | 3.1 (8.5)
Statistical Analysis 1: Comparison: Vericiguat (Baseline) vs Vericiguat Group (Follow-up Visit); The analysis compares the relative change in coronary cross-sectional area (%) from that at rest to that during isometric handgrip exercise in the vericiguat group between that measured at baseline and that measured at six weeks following initiation of titrated dose; Test type: Other — Single group analysis; p = 0.0002, t-test, 2 sided

3. Primary Outcome: Absolute Change in Coronary Cross-sectional Area (in mm²) Between the Vericiguat Group and the Placebo Group as Assessed by Magnetic Resonance Imaging (MRI)
Description: The difference in absolute change in coronary cross-sectional area (in mm²) from rest to isometric handgrip exercise (IHE) as assessed by MRI.
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Population: In the vericiguat arm, two participants withdrew. One withdrew due to personal bereavement following the unexpected death of a close friend, and the other withdrew due to lightheadedness and nausea following alcohol intake.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 21 | 11
mm^2 | 0.40 (1.28) | -0.003 (1.18)
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Other — Two-group analysis; p = 0.528, t-test, 2 sided

4. Primary Outcome: Difference in Percent Change in Coronary Cross-sectional Area (as Percentage) Between the Vericiguat Group and the Placebo Group as Assessed by Magnetic Resonance Imaging (MRI)
Description: The difference in percentage change in coronary cross-sectional area (%) from rest to isometric handgrip exercise (IHE) between the vericiguat and placebo groups, as assessed from the baseline MRI to the follow-up MRI, six weeks following initiation of the titrated dose.
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: % change coronary cross-sectional area
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 21 | 11
% change coronary cross-sectional area | 9.9 (9.80) | 8.8 (13.20)
Statistical Analysis 1: Comparison: Vericiguat vs Placebo; Test type: Other — Multiple linear regression; Regression, Linear — 0.0497; Slope = 6.34

5. Secondary Outcome: Changes in Interleukin 1 (IL-1) Measured Using Blood Samples (in pg/mL)
Description: IL-1 (in pg/mL), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Reporting Status: Not Posted, anticipated posting 2026-07

6. Secondary Outcome: Changes in Interleukin 6 (IL-6) Measured Using Blood Samples (in pg/mL)
Description: IL-6 (in pg/mL), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Reporting Status: Not Posted, anticipated posting 2026-07

7. Secondary Outcome: Changes in Interleukin 10 (IL-10) Measured Using Blood Samples (in pg/mL)
Description: IL-10 (in pg/mL), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Reporting Status: Not Posted, anticipated posting 2026-07

8. Secondary Outcome: Changes in Tumor Necrosis Factor (TNF)-Alpha Measured Using Blood Samples (in pg/mL)
Description: TNF-alpha (in pg/mL), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Reporting Status: Not Posted, anticipated posting 2026-07

9. Secondary Outcome: Changes in High Sensitivity C-Reactive Protein (hsCRP) Measured Using Blood Samples (in mg/L)
Description: hsCRP (in mg/L), an inflammatory marker, will be measured in blood samples to assess changes from baseline.
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Reporting Status: Not Posted, anticipated posting 2026-07

10. Secondary Outcome: Changes in Cyclic Guanosine Monophosphate (cGMP) Measured Using Blood Samples (in Pmol/mL)
Description: cGMP (in pmol/mL), a mediator in the nitric oxide pathway, will be measured in blood samples to assess changes from baseline.
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Reporting Status: Not Posted, anticipated posting 2026-07

11. Secondary Outcome: Changes in Left Ventricular Ejection Fraction (as Percentage) as Assessed by Echocardiography
Description: An ultrasound evaluation of the heart will be performed to assess the impact of vericiguat on left ventricular ejection fraction (%).
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Reporting Status: Not Posted, anticipated posting 2026-07

12. Secondary Outcome: Changes in e' Velocities (in cm/s) as Assessed by Echocardiography
Description: An ultrasound evaluation of the heart will be performed to assess the impact of vericiguat on e' velocities (in cm/s).
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Reporting Status: Not Posted, anticipated posting 2026-07

13. Secondary Outcome: Changes in E/e' Ratio as Assessed by Echocardiography
Description: An ultrasound evaluation of the heart will be performed to assess the impact of vericiguat on the E/e' ratio.
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Reporting Status: Not Posted, anticipated posting 2026-07

14. Secondary Outcome: Changes in Left Atrium Volume Index (in mL/BSA) as Assessed by Echocardiography
Description: An ultrasound evaluation of the heart will be performed to assess the impact of vericiguat on the left atrium volume index (in mL/BSA).
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Reporting Status: Not Posted, anticipated posting 2026-07

15. Secondary Outcome: Changes in Peak Tricuspid Regurgitation (TR) Velocity (in m/s) as Assessed by Echocardiography
Description: An ultrasound evaluation of the heart will be performed to assess the impact of vericiguat on peak TR velocity (in m/s).
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Reporting Status: Not Posted, anticipated posting 2026-07

16. Secondary Outcome: Changes in Strain (as Percentage) as Assessed by Echocardiography
Description: An ultrasound evaluation of the heart will be performed to assess the impact of vericiguat on strain (as percentage).
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Reporting Status: Not Posted, anticipated posting 2026-07

17. Secondary Outcome: Absolute Change in Coronary Flow (in mL/Min) Within the Vericiguat Group as Assessed by Magnetic Resonance Imaging (MRI)
Description: The absolute changes in coronary flow (in mL/min) with isometric handgrip exercise (IHE) in the group randomized to vericiguat from that measured at baseline, prior to the initiation of vericiguat, to that measured at the end of the study drug administration period as assessed by MRI.
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Reporting Status: Not Posted, anticipated posting 2026-07

18. Secondary Outcome: Relative Change in Coronary Flow (as Percentage) Within the Vericiguat Group as Assessed by Magnetic Resonance Imaging (MRI)
Description: The relative changes in coronary flow (as percentage) with isometric handgrip exercise (IHE) in the group randomized to vericiguat from that measured at baseline, prior to the initiation of vericiguat, to that measured at the end of the study drug administration period as assessed by MRI.
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Reporting Status: Not Posted, anticipated posting 2026-07

19. Secondary Outcome: Absolute Change in Coronary Flow (in mL/Min) Between the Vericiguat Group and the Placebo Group as Assessed by Magnetic Resonance Imaging (MRI)
Description: The absolute changes in coronary flow (in mL/min) with isometric handgrip exercise (IHE) in the vericiguat group as compared to the placebo group as assessed by MRI.
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Reporting Status: Not Posted, anticipated posting 2026-07

20. Secondary Outcome: Relative Change in Coronary Flow (as Percentage) Between the Vericiguat Group and the Placebo Group as Assessed by Magnetic Resonance Imaging (MRI)
Description: The relative changes in in coronary flow (as percentage) with isometric handgrip exercise (IHE) in the vericiguat group as compared to the placebo group as assessed by MRI.
Time Frame: Baseline and 6 weeks following initiation of up-titrated dose
Reporting Status: Not Posted, anticipated posting 2026-07

ADVERSE EVENTS:
Time Frame: up to 156 days
Arm/Group | Vericiguat | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/11
Other Adverse Events (participants affected / at risk) | 11/23 | 9/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vericiguat (N=23) | Placebo (N=11)
Orthostatic dizziness (Vascular disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Heartburn (Gastrointestinal disorders) | 3 | 0
Dizziness (General disorders) | 1 | 3
Unsteadiness (General disorders) | 0 | 2
Forgetfulness (Nervous system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting after alcohol consumption (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Syncope (Vascular disorders) | 1 | 0
Palpitations after influenza vaccination (Cardiac disorders) | 0 | 1
Anxiety following mother's cancer diagnosis (Social circumstances) | 1 | 0
Chest discomfort with exercise (Cardiac disorders) | 1 | 0
Epitaxis (General disorders) | 1 | 0
Dry cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased thirst (General disorders) | 0 | 1
Rash following yard work (Skin and subcutaneous tissue disorders) | 0 | 1
Low hemoglobin (Blood and lymphatic system disorders) | 1 | 0
Low fasting glucose (General disorders) | 1 | 1
Low potassium (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT05711719/Prot_SAP_000.pdf